CLINICAL TRIAL: NCT04726254
Title: The JUvaLIfe Registry
Brief Title: The JULI Registry--Hemp and Cannabis Observational Registry
Acronym: JULI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Juva Life (Industry)
Collaborators: Targeted Medical Education (Other)
Responsible Party: Sponsor
Other Study IDs: JULI1000
Record Dates: First submitted 2021-01-24; First posted 2021-01-27 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pain; Appetite Disorders; Neuropathy; Menopausal Syndrome; Anxiety; Sleep Disturbance; Nausea
MeSH Terms: conditions — Chronic Pain; Feeding and Eating Disorders; Anxiety Disorders; Parasomnias; Nausea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The JuLi Registry seeks to fill some of the gaps associated with the clinical use of CBD (cannabidiol) and other cannabinoid formulations including THC and others. The overarching goal of this Registry is to rapidly advance research and understanding of the use of cannabis and hemp-based formulations, in the clinical community setting, when it is utilized to manage the symptoms of cancer treatment and other underlying health issues. These symptoms include nausea, neuropathy, and sleeplessness and chronic pain.

DETAILED DESCRIPTION:
The JuLi Registry seeks to fill some of the gaps associated with the clinical application of CBD (cannabidiol) and other cannabinoid formulations including THC and others. It will also serve as a platform for discovery, whereby observations of patient symptoms, specific cannabis formulations, delivery methods and clinical outcomes, become the source of more in-depth research projects.

The JuLi Registry is a prospective observational Registry documenting utility and patient experience for patients seeking to use therapeutic cannabis and hemp-based products as a means of symptom relief and management related to various diseases.

Targeted symptoms and conditions include:

* Chronic Pain
* Neuropathy
* Sleeplessness
* Poor Appetite
* Nausea
* Anxiety
* Menopausal symptoms

Data to be recorded includes:

* Basic demographics of patients using cannabis-based or hemp-based products
* Disease diagnoses and symptoms for which patients are seeking management
* Cannabinoid formulation, chemical composition, amount (in milligrams), dose and utilization
* Patient Reported Outcomes (PRO) using, where possible, validated measures of sleep, pain, appetite, etc.
* Physician and patient utilization of these data to manage prescription medication recommendations and usage, including discontinuation of opiates or reduction in use of opiates after initiation of cannabis- or hemp-based products
* Overall impact on clinical or patient treatment plan

The purpose of this Registry is to provide a platform for physicians and patients to collaborate on hemp and cannabis research and advance the understanding of the application of cannabinoids for symptom relief associated with various medical conditions.

Patients greater than or equal to 21 years of age seeking to use CBD or other cannabis-based formulations, where legal, will be invited to participate.

Data collected in the normal course of a patient's visit and follow up are entered. This is an observational study; no specific patient interventions are required. Patients must have requested a cannabis-based medicament from their provider. Or be otherwise deemed eligible per the research protocol and choose to participate in a self-directed manner.

Data will be collected at various time points, including:

1. At the time patients first request cannabis or hemp based products
2. At various recommended and voluntary time points, collected via PRO surveys
3. Daily or whenever they are using their products via the use of a study app
4. When patients return to their providers during the course of normal clinical care

All patients must sign an electronic informed consent form prior to their prospective data being entered into the Registry.

All demographic, diagnostic, hemp/cannabis formulation and follow up data will be entered by patients. Consented patients will record compliance with recommendations, usage and symptom relief. They will be asked to take symptom specific surveys.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* Have requested from and/or decided with their providers to try CBD (hemp-based) or other cannabis products to relieve one or more symptoms related to a medical diagnosis
* Consent to have their health data included in a Registry and participate in PRO (patient reported outcomes) surveys and data collection via a study app.

Exclusion Criteria:

* Patient pregnant
* Unwilling or unable to provide informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients greater than or equal to 21 years of age who are seeking to use hemp-based or cannabis-based formulations to relieve symptoms associated with medical interventions or conditions
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Symptom Relief | 3 months
  Percentage of patients who obtain and report symptom relief, by symptom, condition and cannabis formulation
Reduction in reliance on Rx medications | 3 months
  Percentage of patients who report reduction or increase in use of Rx medications

SECONDARY OUTCOMES:
Reduction in reliance on OTC medications | 3 months
  Percentage of patients who report reduction or increase in use of Rx medications

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Precision Cancer Specialists, Los Gatos, California
  - Justin Lo MD, San Jose, California
  - Nashville Breast Center, Nashville, Tennessee
  - Dallas Surgical Group, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zou S, Kumar U. Cannabinoid Receptors and the Endocannabinoid System: Signaling and Function in the Central Nervous System. Int J Mol Sci. 2018 Mar 13;19(3):833. doi: 10.3390/ijms19030833. PMID 29533978
- [Result] Freitas HR, Isaac AR, Malcher-Lopes R, Diaz BL, Trevenzoli IH, De Melo Reis RA. Polyunsaturated fatty acids and endocannabinoids in health and disease. Nutr Neurosci. 2018 Dec;21(10):695-714. doi: 10.1080/1028415X.2017.1347373. Epub 2017 Jul 7. PMID 28686542